CLINICAL TRIAL: NCT04703920
Title: A Phase 1 Dose-Escalation Trial of Talazoparib in Combination With Belinostat for Metastatic Breast Cancer, Metastatic Castration Resistant Prostate Cancer, and Metastatic Ovarian Cancer
Brief Title: Talazoparib in Combination With Belinostat for Metastatic Breast Cancer, Metastatic Castration Resistant Prostate Cancer, and Metastatic Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Pfizer (Industry); Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2020.122; HUM00187603 (Other: University of Michigan)
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer; Metastatic Castration-resistant Prostate Cancer; Metastatic Ovarian Carcinoma; Metastic or Unresectable Pancreatic Adenocarcinoma
Keywords: PARP inhibitor
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — talazoparib; belinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Talozoparib in combination with Belinostat (Experimental): Patients will receive Talozoparib in combination with Belinostat
  Interventions: Drug: Talazoparib; Drug: Belinostat

INTERVENTIONS:
Drug: Talazoparib — Talazoparib will be administered in increasing doses up to 1 mg orally once a day.
Drug: Belinostat — Belinostat will be administered in increasing doses up to 1000 mg/m2 IV once daily on days 1-5 of a 21-day cycle.

SUMMARY:
This Phase 1 dose-escalation trial is to determine the safety, tolerability and recommended phase 2 dose of talazoparib in combination with belinostat in subjects with Metastatic Breast Cancer, Metastatic Castration Resistant Prostate Cancer, and Metastatic Ovarian Cancer.

ELIGIBILITY:
Inclusion Criteria:

* One of the following disease types: Men or women with histologically confirmed metastatic or unresectable breast cancer that is HER2 negative as assessed by 2018 ASCO-CAP guidelines. Trial participants with hormone receptor positive disease must have progression on at least one hormonal therapy and a CDK inhibitor AND be considered a candidate for chemotherapy; OR, Men with metastatic castration resistant prostate cancer with progression on androgen deprivation therapy and at least one additional agent in the metastatic setting; OR, Women with metastatic high grade serous ovarian cancer with progression on at least one chemotherapy agent; OR, men or women with metastatic or unresectable pancreatic adenocarcinoma with progression on at least one chemotherapy regimen in the metastatic/unresectable setting
* Measurable disease as defined by RECIST 1.1 criteria.
* Trial participants must be at least 21 days from last dose of chemotherapy and recovered from all chemotherapy-related reversible toxicity to Grade 0 or 1, with the exception of alopecia and neuropathy.
* The last radiation therapy (including palliative radiation) must have occurred ≥3 weeks prior to study registration.
* Trial participants must have experienced disease progression at the time of study enrollment.
* ECOG performance status of 0 or 1.
* Adequate organ and marrow function per protocol.
* Trial participants with treated brain metastases are eligible provided the metastases are recently treated and/or clinically stable and greater than 4 weeks has elapsed from time of treatment and date of initiation of study drug.
* Trial participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen should be included.
* Males and females of reproductive potential must use two forms of effective contraception during the duration of the trial and for minimum of 7 months after last dose of study drug. A woman of reproductive potential is defined as a premenopausal female with intact uterus and ovaries. For women, non-childbearing potential is defined as:

  * ≥45 years of age and has not had menses for >2 years.
  * Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation.
  * Post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Previous or current treatment with a histone deacetylase inhibitor (HDACi)S.
* Participation in other investigational studies concurrently if these therapies include a therapeutic intervention.
* Treatment with any investigational agent within 30 days (or 5 serum half-lives of the investigational drug, whichever is longer) of enrollment.
* Evidence of current serious uncontrolled concomitant cardiovascular nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator, including, but not limited to:

  * Myocardial infarction or arterial thromboembolic events within 6 months prior to screening or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a QTc interval > 450 msec.
  * Uncontrolled hypertension or diabetes mellitus.
  * Another known malignancy that is progressing or requires active treatment.
  * Active infection requiring systemic therapy.
  * Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
* Allergy to talazoparib, belinostat or to the inactive components of talazoparib or belinostat formulations.
* Pregnancy or breastfeeding.
* QTc ≥ 450 ms or congenital long QT syndrome given potential for prolongation with belinostat.
* Current or anticipated use within 7 days prior to enrollment, or anticipated use during the study of drugs which are moderate or strong inhibitors of UGT1A1 per protocol.
* Current or anticipated use within 7 days prior to enrollment, or anticipated use during the study, of strong P-gp inhibitors per protocol.
* Subjects homozygous for UGT1A1*28 allele; this will be determined via clinical testing by polymerase chain reaction with capillary electrophoresis by the University of Michigan Molecular Diagnostics laboratory.
* Any medical or psychological condition that in the opinion of the principal investigator would interfere with safe completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) within the first two cycles of treatment | 10 weeks
  Number of DLT's experienced by participants within the first two cycles. A DLT will be defined as any treatment related toxicity of grade 3 or 4 unless otherwise defined in the protocol. DLTs will be assessed via the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Proportion of patients experiencing toxicities. Participants may continue to receive the investigational study therapy until disease progression or unacceptable toxicity. | Up to 30 days post last treatment, up to approximately 6 months
  The proportion of patients experiencing toxicities will be reported by dose level and grade. Toxicities and grading per the NCI CTCAE version 5.0.
Plasma concentrations of talazoparib at steady state | Day 5 of cycle 1; up to day 5 of cycle 3
  Plasma concentrations of talazoparib at steady state will be measured to evaluate its pharmacokinetic (PK) profile, with combination therapy of talazoparib and belinostat. Sparse PK assessment will occur at multiple time points from day 5 of cycle 1 through day 5 of cycle 3 in order to assess steady-state trough levels. The plasma concentrations will be determined by liquid chromatography, high-resolution mass spectrometry, and summarized descriptively by dose level.
Plasma concentrations of belinostat at steady state | Day 5 of cycle 1; up to day 5 of cycle 3
  Plasma concentrations of belinostat at steady state will be measured to evaluate its PK profile, with combination of talazoparib and belinostat. Sparse PK assessment will occur at multiple time points from day 5 of cycle 1 through day 5 of cycle 3 in order to assess steady-state trough levels. The plasma concentrations will be determined by liquid chromatography, high-resolution mass spectrometry, and summarized descriptively by dose level.
Number of patients with an objective response | Up to 30 days post last treatment, up to approximately 6 months
  Number of patients with an objective response per the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 will be reported by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Burness, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No